CLINICAL TRIAL: NCT03946280
Title: Utility of 3D Navigation to Reduce Ionizing Radiation in Common Flutter Ablation. Study of Personnel and Patient Dosimetry
Acronym: DOSIMETRY-AFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DOSIMETRY - FLUTTER
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Auricular Flutter; Radiation Exposure
Keywords: ALARA; radiation exposure; Flutter ablation
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Intervention Model Description: Randomized study, patients are allocated to 1 of the 2 groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopy Group (Other): Patient undergoing common flutter (AFL) ablation procedure using conventional X-ray based fluoroscopy for for catheter tracking
  Interventions: Procedure: conventional X-ray based Fluoroscopy
- 3D Group (Experimental): Patient undergoing common flutter (AFL) ablation procedure using the low X-ray 3D navigation technique for for catheter tracking
  Interventions: Procedure: low X-ray 3D navigation technique

INTERVENTIONS:
Procedure: conventional X-ray based Fluoroscopy — catheter tracking via conventional X-ray based Fluoroscopy
  Arms: Fluoroscopy Group
Procedure: low X-ray 3D navigation technique — catheter tracking via low X-ray 3D navigation technique
  Arms: 3D Group

SUMMARY:
Common Flutter ablation technique use low X-ray based three-dimension (3D) navigation for catheter tracking, have become a popular implementation to treat patient's underlying arrhythmia. Compared with fluoroscopy, the gold standard X-ray based method, this recent technique provides the required anatomical information and reduce risk associated with ionizing radiation exposure. Besides Practical Guidelines "as low as reasonably achievable (ALARA) to minimize and normalize radiation exposure had been published so far. The risk of developing acute radiation associated injuries still remains high. In the present study we will compare two groups of patients undergoing into cavotricuspid isthmus (CTI) ablation using either the 3D navigation ("Ensite NavX system") (n = 25) or conventional fluoroscopy (n = 25). Further developing the 3D navigation technique will help to increase safety during the treatment, for both patients and the personnel and increase the success rate during the electrophysiological (EP) interventional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Sick adult patients with Atrial Flutter arrythmia
* patients able to consent.
* patients scheduled to receive cavotricuspid isthmus ablation treatment

Exclusion Criteria:

* patients who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants | through study completion, an average of 2 year
  two groups and 25 patiens within each group
age | at the moment the patient was recruited for the study
  age in years of every patient in the study
Electrophysiology procedure time (EP time) | at the moment of the intervention
  time the intervention last in minutes
Radiofrecuency ablation time | at the moment of the intervention
  time radiofrecuency are applied within the EP time in minutes/ seconds
Total Fluoroscopy time | at the moment of the intervention
  time the patiens receive x ray radiation along the intervention in minutes/ seconds
Time without fluoroscopy | at the moment of the intervention
  time the patiens do not receive any x ray radiation along the intervention in minutes/ seconds
Dose area product | at the moment of the intervention
  Global Radiation dose emited by the x-ray tube in mgcm2
Radiation dose TLD in patient (5 TLD) | at the moment of the intervention
  five thermoluminescent dosimeters are placed on the body of the patient in mgcm2
Radiation dose TLD in operator (3 TLD) | at the moment of the intervention
  three thermoluminescent dosimeters are placed on the body of the patient in mgcm2
readmission | within 12 months following the EP
  times the patient is readmitted in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Scavée, PhD, Principal Investigator — Cliniques Universitaires St Luc
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No